CLINICAL TRIAL: NCT04403555
Title: The Efficacy of Ivermectin in COVID-19 Treatment
Brief Title: Ivermectin as a Novel Therapy in COVID-19 Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tanta covid treatment
Record Dates: First submitted 2020-05-23; First posted 2020-05-27 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: COVID
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin (Experimental): Ivermectin plus standard of care treatment Dose 2 tablets 12mg per day for 3 days
  Interventions: Drug: Ivermectin
- Standard of care (No Intervention): Standard of care treatment

INTERVENTIONS:
Drug: Ivermectin — Ivermectin treatment
  Other Names: iverzine, ivermectin
  Arms: Ivermectin

SUMMARY:
Efficacy of Ivermectin in COVID-19 treatment

DETAILED DESCRIPTION:
Clinical Study Evaluating the Efficacy of Ivermectin in COVID-19 treatment

ELIGIBILITY:
Inclusion Criteria:

* All Adult Patients aging from 20 to 65 years-old with COVID-19 confirmed by pharyngeal swab PCR.

Exclusion Criteria:

* Allergy or contraindication to the drugs used in the study.
* Pregnant and lactating mothers.
* Patients with cardiac problems.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
The number of patients with mortality | 1 month
  Improvement of survival

SECONDARY OUTCOMES:
Length of hospital stay | 1 month
  Effect on the length of hospital stay
The need for mechanical ventilation | 1 month
  Need for mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: sherief Abd-Elsalam, Ass. Prof., Principal Investigator — ass. Prof. Tropical Medicine
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No